CLINICAL TRIAL: NCT03210025
Title: Clinical Bioequivalence Study on Two Methyldopa Tablet 250mg Formulations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bright Future Pharmaceuticals Factory O/B Bright Future Pharmaceutical Laboratories Limited (Industry)
Collaborators: Chinese University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: BABE-P15-096
Record Dates: First submitted 2017-07-03; First posted 2017-07-06 (Actual); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Healthy
MeSH Terms: interventions — Tablets; Methyldopa

STUDY DESIGN:
Intervention Model Description: Single-dose, two-treatment, two-period, two-sequence crossover
Masking Description: Open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BF-Methyldopa Tablet 250mg (Experimental): During the study session, healthy subjects will be administered a single dose of BF-Methyldopa Tablet 250mg after an overnight fast of approximately 10 hours
  Interventions: Drug: BF-Methyldopa 250mg Tablet
- Metopa Tab 250mg (Active Comparator): During the study session, healthy subjects administered a single dose of Metopa Tablet 250mg after an overnight fast of approximately 10 hours
  Interventions: Drug: Metopa Tab 250mg

INTERVENTIONS:
Drug: BF-Methyldopa 250mg Tablet — BF-Methyldopa 250mg Tablet is a generic product manufactured by Bright Future Pharmaceuticals Factory O/B Bright Future Pharmaceutical Laboratories Limited
  Other Names: Methyldopa 250mg Tablet
  Arms: BF-Methyldopa Tablet 250mg
Drug: Metopa Tab 250mg — Metopa Tab 250mg is manufactured by APT
  Other Names: Methyldopa 250mg Tablet
  Arms: Metopa Tab 250mg

SUMMARY:
The objective of the study is to compare the bioavailability of a generic product of methyldopa with that of a reference product when administered to healthy volunteers under fasting condition. The test product is BF-Methyldopa Tablet 250mg (HK Reg. No. HK-62917) manufactured by Bright Future Pharmaceuticals Factory O/B Bright Future Pharmaceutical Laboratories Limited, and the reference product is Metopa Tab 250mg (HK Reg. No. HK-44620). The plasma pharmacokinetic data of Methyldopa obtained from two formulations will be used to access the interchangeability of the products.

DETAILED DESCRIPTION:
It is planned to enroll 16 to 30 healthy subjects, with an aim to obtain at least 12 evaluable subjects. The study design is a single-dose, two-treatment, two-period, two-sequence crossover with a washout period of one to two weeks. During each study session, the subjects will be administered a single oral dose of 250mg methyldopa (one BF-Methyldopa Tablet 250mg or one Metopa Tab 250mg) after an overnight fast of approximately 10 hours. Venous blood samples will be collected at pre-dose (0h) and at 0.75 (45min), 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12 and 24 hours post-dose. The plasma concentrations of methyldopa will be determined by a validated assay. The non-compartmental method will be used to analyze the plasma concentration-time data and calculate the main pharmacokinetic parameters such as Cmax, Tmax, AUC0-last, AUC0-inf, and T1/2. Anylasis of variance (ANOVA) will be conducted on logarithmically transformed Cmax, AUC0-last and AUC0-inf using the General Linear Model. The two one-side tests will be used to calculate the 90% confidence intervals for the mean difference in AUC0-last, AUC0-inf and Cmax and to assess the bioequivalence of the two products.

ELIGIBILITY:
Inclusion Criteria:

* Male and non-pregnant female, 18 to 55 years of age
* Body Mass Index between 18 to 27 kg/m2
* Accessible vein for blood sampling
* High probability for compliance and completion of the study
* Female subjects must agree to practice abstinence or take effective contraceptive methods to prevent pregnancy from the start of screening until two weeks of last dose administration.

Exclusion Criteria:

* Clinical significant hepatic, renal, biliary, cardiovascular, gastrointestinal, haematological and other chronic and acute diseases within 3 months prior to the study
* Clinical significant abnormality in physical examination, vital signs, ECG evaluation, urine test, blood chemistry or haematological test
* Tobacco use in any forms
* Regular consumer of alcohol
* Blood donation within 4 weeks prior to the start of the study
* Use of Methyldopa within 4 weeks before the study
* Use of antihypertensive medications within 4 weeks before the study
* Volunteer in any other clinical drug study within 2 months prior to this study
* Hypersensitivity to Methyldopa or other drugs in its class
* History of drug abuse in any form
* Female subjects who are breastfeeding or pregnant.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2017-09-20 (Actual); Primary Completion 2017-10-15 (Actual); Study Completion 2017-10-15 (Actual)

PRIMARY OUTCOMES:
Cmax of Methyldopa | 24 hours
AUC of Methyldopa | 24 hours

SECONDARY OUTCOMES:
Tmax of Methyldopa | 24 hours
Elimination half-life (t1/2) of Methyldopa | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Zhong Zuo, Principal Investigator — School of Pharmacy, The Chinese University of Hong Kong; Riza Ozaki, Study Director — Phase 1 Clinical Trial Centre, The Chinese University of Hong Kong; Brian Tomlinsion, Study Director — Department of Medicine and Therapeutics, The Chinese University of Hong Kong
Locations (1):
- Phase 1 Clinical Trial Centre, The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided